CLINICAL TRIAL: NCT02248129
Title: Pharmaco-epidemiological Study Describing a Population of Hypertensive Patients Treated in General Practice With a Fixed-dose Combination of Telmisartan and Hydrochlorothiazide, the Level of Blood Pressure Control and the Modalities of Arterial Hypertension Management
Brief Title: Pharmaco-epidemiological Study Describing a Population of Hypertensive Patients Treated With a Fixed-dose Combination of Telmisartan and Hydrochlorothiazide
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 502.508
Record Dates: First submitted 2014-09-22; First posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — telmisartan, hydrochlorothiazide drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Hypertensive patients
  Interventions: Drug: Telmisartan and hydrochlorothiazide

INTERVENTIONS:
Drug: Telmisartan and hydrochlorothiazide

SUMMARY:
Study to compare the level of blood pressure control in hypertensive, hypertensive diabetics and hypertensive with renal insufficiency (observed data) in the study population, with the objectives of the High Authority for Health recommendations (benchmark)

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive patients already treated for at least 1 month with Telmisartan plus hydrochlorothiazide, consulting the physician consecutively for whatever reason

Exclusion Criteria:

* NA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hypertensive patients treated in general practice
Sampling Method: Non-Probability Sample
Enrollment: 4255 (Actual)
Dates: Start 2006-04; Primary Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with low blood pressure | up to 4 weeks
  lower than 140/90 mmHg in the general population of hypertensive patients, hypertensive diabetics and hypertensive with renal insufficiency

SECONDARY OUTCOMES:
Number of patients with adverse events | up to 4 weeks